CLINICAL TRIAL: NCT04835103
Title: Build a Psychosomatic Research Clinic for Providing Comprehensive Managements to Somatoform Patients
Brief Title: Build a Research Clinic for Somatoform Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201812052RIND
Record Dates: First submitted 2021-01-29; First posted 2021-04-08 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2023-12

CONDITIONS: Somatoform Disorders; Somatic Symptom Disorder
Keywords: somatoform disorders; somatic symptom disorder; psychosomatic medicine; medically unexplained symptoms
MeSH Terms: conditions — Somatoform Disorders; Medically Unexplained Symptoms

STUDY DESIGN:
Intervention Model Description: Case management, a case manager will actively contact and follow the patient's physical and psychological conditions, and provide disease-specific psychoeducation; psychotherapy for patients with somatoform disorders (combined cognitive-behavioral treatment and biofeedback therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Set a case management model for somatoform patients (Other): Somatoform patients receiving case management, single group assignment, open label
  Interventions: Behavioral: CM
- Time-limited psychotherapy for somatoform patients (Other): Somatoform patients receiving psychotherapy (based on cognitive-behavioral therapy and biofeedback therapy) vs treatment as usual, open label, non-randomized
  Interventions: Behavioral: P/T

INTERVENTIONS:
Behavioral: CM — Case management, a case manager will actively contact and follow the patient's physical and psychological conditions, and provide disease-specific psychoeducation
  Arms: Set a case management model for somatoform patients
Behavioral: P/T — Psychotherapy, based on both cognitive-behavioral therapy and biofeedback therapy, structuralized, 6-10 sessions, performed by a psychiatrist or psychologist
  Arms: Time-limited psychotherapy for somatoform patients

SUMMARY:
To investigate the effects of the two following interventions on somatoform patients:1. case management model2. psychotherapy, based on cognitive-behavioral therapy and biofeedback therapy

DETAILED DESCRIPTION:
Patients with presentations of somatic symptoms and associated psychological features are named as "somatoform disorders" in psychiatric field. Because the patients' concerns are somatic distress, they often seek help in non-psychiatric clinics. However, the symptoms are usually medically unexplained. This group of diagnoses can be managed from the psychiatric perspective, including medications and psychotherapies. However, many patients do not receive psychiatric management in current medical practice. The goal of this project is to establish an association named "psychosomatic center" for providing comprehensive evaluations and treatments to the somatoform patients. Besides the psychiatrist, a case manager, a clinical psychologist, and a research assistant will be included in this association for the purposes of connection, performing psychotherapy and examinations. After entering the psychosomatic clinic, the investigators will routinely perform diagnostic interview, measure psychological and physiological features, and arrange individualized treatment program. The investigators will follow the important psychological and biological indexes every 3-6 months for building a cohort. At the same time, the case manager will connect with non-psychiatric clinics for ensuring the patients physical problems to be managed. The investigators expect this project to enhance the quality of treatment on the patients, to reduce the excessive examinations for the frequent attenders, and to improve the emotional burden of medical staffs.

ELIGIBILITY:
Inclusion Criteria:

* 1. Between 15 and 80 years old
* 2. Meet the diagnosis of DSM-5 somatic symptom disorder

Exclusion Criteria:

* 1. With psychotic symptoms (such as schizophrenia, bipolar disorder with psychotic symptoms) or cognitive impairment
* 2. Having potentially lethal physical diseases (such as cancer, coronary artery diseases, cerebrovascular diseases; because under this condition, high health anxiety is quite rational. Patients with common physical diseases can still enter this trial)
* 3. Unable to read or understand the questionnaires

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Patient Health Questionnaire-15 (PHQ-15) score at 3 months and 6 months (for psychotherapy); changes from baseline PHQ-15 score at 3, 6, 12, 24 months (for case management) | 3, 6 months after initiating psychotherapy (for psychotherapy); 3, 6, 12, 24 months after initiating case management (for case management)
  PHQ-15 is a scale rating the severity of somatic distress. It is a 3-point Likert scale with 15 items. The scores range from 0 (lowest level of somatic distress) to 30 (highest level of somatic distress).
Changes from baseline Health Anxiety Questionnaire (HAQ) score at 3 months and 6 months (for psychotherapy); changes from baseline HAQ score at 3, 6, 12, 24 months (for case management) | 3, 6 months after initiating psychotherapy (for psychotherapy); 3, 6, 12, 24 months after initiating case management (for case management)
  HAQ is a scale rating the severity of health anxiety. It is a 4-point Likert scale with 21 items. The scores range from 0 (lowest level of health anxiety) to 63 (highest level of health anxiety).

SECONDARY OUTCOMES:
Scores of Scale for the Assessment of Illness Behavior (SAIB) | 3, 6, 12, 24 months
  SAIB is a scale rating the illness behavior. It is a 4-point Likert scale with 25 items. The scores range from 0 to 75.
Scores of Cognition About Body and Health Questionnaire (CABAH) | 3, 6, 12, 24 months
  CABAH is a scale rating the cognition about health anxiety. It is a 4-point Likert scale with 39 items. The scores range from 0 to 117.
Scores of Beck Depression Inventory-II (BDI- II) | 3, 6, 12, 24 months
  BDI- II is a scale rating the severity of depression. It is a 4-point Likert scale with 21 items. The scores range from 0 (lowest level of depression) to 63 (highest level of depression).
Scores of Beck Anxiety Inventory (BAI) | 3, 6, 12, 24 months
  BAI- II is a scale rating the severity of anxiety. It is a 4-point Likert scale with 21 items. The scores range from 0 (lowest level of anxiety) to 63 (highest level of anxiety).
Penn State Worry Questionnaire (PSWQ) | 3, 6, 12, 24 months
  PSWQ-16 is a scale rating the severity of worry. It is 5-point Likert scale with 16 items. The scores range from 1 (lowest level of worry) to 80 (highest level of worry).
Scores of WHOQOL-BREF | 3, 6, 12, 24 months
  It is a self-report questionnaire measuring health-related quality of life. It is a 4-point Likert scale with 28 items, which belong to 5 domains (the overall, physical, psychological, social and environmental domains). The scores of each domain are usually normalized with 0-20 or 0-100.
Changes from baseline standard deviation of normal to normal RR intervals (SDNN) | 3, 6, 12, 24 months
  SDNN reflects all the cyclic components responsible for variability in the period of recording, therefore it represents total variability.
Changes from baseline high-frequency power (HF) | 3, 6, 12, 24 months
  HF component of HRV represents parasympathetic activity.
Changes from baseline ratio of low-frequency power to high-frequency power (LF/HF) | 3, 6, 12, 24 months
  LF/HF was considered to reflect sympathovagal balance by some scholars.
Changes from baseline value of skin conductance. | 3, 6, 12, 24 months
  In skin conductance, an electrodermograph imposes an imperceptible current across the skin and measures how easily it travels through the skin. Skin conductance is usually considered as a biomarker of sympathetic activity.
Changes from baseline value of Respiratory sinus arrhythmia | 3, 6, 12, 24 months
  Respiratory sinus arrhythmia is an index combining the heart rate and respiratory signal, it represents parasympathetic activity.
Changes from baseline value of Finger temperature. | 3, 6, 12, 24 months
  Finger temperature is found to be related to emotional disturbance (such as depression and anxiety), and it is often used in biofeedback therapy.
Changes from baseline value of electromyogram | 3, 6, 12, 24 months
  Electromyogram is found to be related to emotional disturbance (such as depression and anxiety), and it is often used in biofeedback therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital Yunlin Branch, Douliu, Taiwan